CLINICAL TRIAL: NCT06569927
Title: Application and Effectiveness of the Perioperative Position Management Based on the ADDIE Model in Patients With Congenital Microtia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FNF202312
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Congenital Microtia
Keywords: Congenital microtia; Position management
MeSH Terms: conditions — Congenital Microtia

STUDY DESIGN:
Intervention Model Description: Subjects were grouped based on admission time to avoid contamination between groups, with data collection for the intervention group conducted after the control group.
Who Masked: Participant
Masking Description: The intervention study used a single-blind design, blinded the subjects, and the patients did not know the specific intervention measures, and did not know whether they were included in the control group or the intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group implemented a perioperative position management program for congenital microtia based on the ADDIE model, in addition to routine position care.
  Interventions: Procedure: Utilization of a perioperative position management protocol for congenital microtia patients based on the ADDIE model.
- Control Group (No Intervention): The control group received routine position care, which included perioperative verbal emphasis on the importance of position by nurses, intraoperative use of hydrocolloid positioning pads to prevent pressure injuries, postoperative nurse monitoring and encouragement of proper positioning, assistance with bed mobility, and guidance on safe ambulation techniques.

INTERVENTIONS:
Procedure: Utilization of a perioperative position management protocol for congenital microtia patients based on the ADDIE model. — Key elements included formation of a multidisciplinary team，perioperative postural management, preoperative sleeping posture adaptability training, neck movement training, standardization of head position angles and head suspension time during surgery, use of protective headrests, attention to transfer and handover procedures, and specially designed pillows.
  Arms: Intervention group

SUMMARY:
Aims and objectives: To evaluate the clinical application and effectiveness of a perioperative position management program constructed using the ADDIE model for patients with congenital microtia.

Background: The primary challenge in auricular reconstruction is the fragility of the reconstructed ear structure, necessitating strict avoidance of postoperative pressure to ensure the surgery's effect. Clinically, this has been found to cause anxiety in patients and their families. Some patients maintain a fixed position to avoid pressure on the reconstructed ear, which may lead to restricted neck movement and a high risk of pressure-related injuries. Therefore, a systematic perioperative position management program for patients with congenital microtia is necessary.

Methods: A quasi-trial design with non-randomized grouping was adopted. Using convenience sampling, 98 patients with congenital microtia admitted to a tertiary specialized hospital in Shanghai from May to August 2023 were included in the control group and received routine care. From September to December 2023, another 98 patients were included in the intervention group, receiving a perioperative position management program in addition to routine care. Effectiveness was evaluated using the Ear Reconstruction Effectiveness Scale, SCARED, Quality of Life Scale for Congenital External and Middle Ear Malformation Patients, SAS, Northwick Park Neck Pain Questionnaire, and Position Execution Checklist.

DETAILED DESCRIPTION:
Auricular reconstruction remains one of the most challenging surgeries due to its delicate structures and potential complications. The reconstructed auricle is too fragile to withstand excessive pressure that will cause blood circulation disturbances or even necrosis. Clinical observations have noted that patients and their families often experience anxiety due to concerns over complications and the impact on recovery, affecting their quality of life. Furthermore, patients frequently hold their heads in a fixed position to prevent pressure on the reconstructed auricle, which results in neck stiffness, asymmetry, and limited mobility. Therefore, effective perioperative position management is crucial for improving surgical outcomes and patient prognosis and alleviating negative emotions in patients and their families.

In our study, we evaluated the clinical usefulness of a perioperative position management program designed using the ADDIE model for patients with microtia. The patients were divided into the experimental group（98 cases）and control group （98 cases）in a quasi-experimental design that used non-randomized grouping. The experimental group received the perioperative position management program in addition to routine care. Key elements included perioperative postural management, preoperative sleeping posture adaptability training, neck movement training, standardization of head position angles and head suspension time during surgery, use of protective headrests, attention to transfer and handover procedures, and specially designed pillows.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital microtia according to the "Chinese Plastic Surgery" criteria, and undergoing ear reconstruction.
* No other severe comorbidities.

Exclusion Criteria:

* Abnormal coagulation function.
* Presence of eczema or infection on the affected side.
* Severe cognitive impairment or mental illness.
* Patient or family disagrees with the study.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Ear Reconstruction Effectiveness Scale | 3 months postoperatively.
  Evaluation was conducted using the surgical outcome scoring system developed by Wei Lü. The scale includes five aspects: (1) The size, position, and realism of the reconstructed ear compared to the healthy side (total score 24 points). (2) The angle size and stability of the cranioauricular angle of the reconstructed ear (total score 12 points). (3) The color of the skin of the reconstructed ear and its coordination with the surrounding skin (total score 10 points). (4) The condition of the local scars at the incision behind the ear (total score 9 points). (5) The presentation of the subunit structure of the reconstructed ear (total score 45 points). A total score greater than 85 is rated as excellent; 75-84 is rated as good; 65-74 is rated as fair; and less than 65 is rated as poor. The specific method of use involves plastic surgeons scoring based on the structure of the child's healthy side or the structure of a normal person's auricle.
Incidence of skin and flap-related complications after ear reconstruction | 3 months postoperatively.
  The researchers independently designed the position execution checklist based on a review of relevant literature. The checklist consists of two parts: (1) Demographic Information: This includes gender, age, education level, and caregivers. (2)Disease-Related Information: This includes the duration of surgery, the side of the surgery, the name of the surgery, instances of reconstructed ear compression, the time period during which the compression occurred, the occurrence of complications, and medication usage.

SECONDARY OUTCOMES:
Quality of Life Scale for Congenital External and Middle Ear Malformation Patients | Within 24 hours prior to discharge.
  This scale is used to assess the quality of life of patients with congenital middle and outer ear deformities, encompassing three dimensions: physical function, psychological state, and social relationships, with a total of 18 items. Each item is rated on a five-point scale from 0 to 4, with a total score ranging from 0 to 80. The higher the score, the poorer the quality of life.
Northwick Park Neck Pain Questionnaire (NPQ) | Within 24 hours prior to discharge.
  This scale is used to assess the function of clinical neck pain patients and consists of 9 items, including pain severity, duration of symptoms, nighttime prickling or numbness, the impact of pain on sleep, social activities, reading, work or household tasks, and driving. If the subject has no driving experience, this item is not scored. Each item is rated on a five-point scale from 0 to 4, with a total score ranging from 0 to 36. The higher the score, the more severe the neck pain.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Within 24 hours prior to discharge.
  This scale is used for self-assessment of anxiety disorders in children and adolescents aged 8-16. It includes five factors: somatization/panic, generalized anxiety, separation anxiety, social phobia, and school phobia, with a total of 41 items. Each item is scored on a three-point scale from 0 to 2. 0: no problem; 1: sometimes; 2: often. The higher the score, the more severe the anxiety.
Self-Rating Anxiety Scale (SAS) | Within 24 hours prior to discharge.
  This scale is used to assess subjective feelings of anxiety and consists of 20 items. Each item is scored on a four-point scale. Five items (items 5, 9, 13, 17, 19) are positively worded, while the remaining 15 items are negatively worded. Patients' families use the Self-Rating Anxiety Scale (SAS) for evaluation, with scores interpreted as follows: less than 50 indicates no anxiety, 50-59 indicates mild anxiety, 60-69 indicates moderate anxiety, and greater than 69 indicates severe anxiety. Higher scores reflect more severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abuhassna, H., Alnawajha, S., Awae, F., Adnan, M., & Edwards, B. (2024). Synthesizing technology integration within the Addie model for instructional design: A comprehensive systematic literature review. Journal of Autonomous Intelligence, 7(5), 1-28. https://doi.org/https://doi.org/10.32629/jai.v7i5.1546
- [Background] Ayhan H, Tastan S, Iyigun E, Ozturk E, Yildiz R, Gorgulu S. The Effectiveness of Neck Stretching Exercises Following Total Thyroidectomy on Reducing Neck Pain and Disability: A Randomized Controlled Trial. Worldviews Evid Based Nurs. 2016 Jun;13(3):224-31. doi: 10.1111/wvn.12136. Epub 2016 Jan 15. PMID 26773539
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Chen X, Ma J, Zhang T. Genetics and Epigenetics in the Genesis and Development of Microtia. J Craniofac Surg. 2024 Feb 12;35(3):e261-6. doi: 10.1097/SCS.0000000000010004. Online ahead of print. PMID 38345940
- [Background] Chen X, Zhang R, Zhang Q, Xu Z, Xu F, Li D, Li Y. Microtia Part II: Post-Operation and Complications Management Lessons from 1012 Ear Reconstruction Operations. Aesthetic Plast Surg. 2022 Dec;46(6):2790-2796. doi: 10.1007/s00266-022-03010-6. Epub 2022 Jul 14. PMID 35835875
- [Background] Deng K, Dai L, Yi L, Deng C, Li X, Zhu J. Epidemiologic characteristics and time trend in the prevalence of anotia and microtia in China. Birth Defects Res A Clin Mol Teratol. 2016 Feb;106(2):88-94. doi: 10.1002/bdra.23462. Epub 2015 Dec 17. PMID 26681129
- [Background] Fan Y, Liu W, Fan X, Niu X, Chen X. Psychosocial status of patients with unilateral and bilateral microtia before auricular reconstruction surgery. Int J Pediatr Otorhinolaryngol. 2021 Dec;151:110928. doi: 10.1016/j.ijporl.2021.110928. Epub 2021 Sep 25. PMID 34607045
- [Background] Han SE, Oh KS. Satisfactory surgical option for cartilage graft absorption in microtia reconstruction. J Craniomaxillofac Surg. 2016 Apr;44(4):471-8. doi: 10.1016/j.jcms.2015.12.015. Epub 2016 Jan 6. PMID 26857756
- [Background] Li H, Wang Y, Qian J, Wang B, Liu T, Zhang Q. A Two-Stage Method for Adult Congenital Microtia: The Essentials of 15-Year Experience. Laryngoscope. 2023 Sep;133(9):2148-2153. doi: 10.1002/lary.30531. Epub 2022 Dec 20. PMID 36537375
- [Background] Li Q, Zhou X, Wang Y, Qian J, Zhang Q. Auricular reconstruction of congenital microtia by using the modified Nagata method: Personal 10-Year experience with 1350 cases. J Plast Reconstr Aesthet Surg. 2018 Oct;71(10):1462-1468. doi: 10.1016/j.bjps.2018.05.036. Epub 2018 Jun 19. PMID 30097399
- [Background] Nuyen BA, Kandathil CK, Saltychev M, Firmin F, Most SP, Truong MT. The Social Perception of Microtia and Auricular Reconstruction. Laryngoscope. 2021 Jan;131(1):195-200. doi: 10.1002/lary.28619. Epub 2020 Apr 10. PMID 32275329
- [Background] Patel KR, Benchetrit L, Ronner EA, Occhiogrosso J, Hadlock T, Shaye D, Quesnel AM, Cohen MS. Development of an interdisciplinary microtia-atresia care model: A single-center 20-year experience. Laryngoscope Investig Otolaryngol. 2022 Nov 16;7(6):2103-2111. doi: 10.1002/lio2.896. eCollection 2022 Dec. PMID 36544952
- [Background] Sevillano-Jimenez A, Romero-Saldana M, Molina-Recio G. Nursing role on rapid recovery programmes fast-track. Enferm Clin (Engl Ed). 2017 Jul 27:S1130-8621(17)30098-0. doi: 10.1016/j.enfcli.2017.06.002. Online ahead of print. English, Spanish. PMID 28757097
- [Background] Turhan Damar H, Ogce Aktas F. Anxiety, Depression, Stress, and Self-Esteem in Turkish Parents of Children with Microtia. Cleft Palate Craniofac J. 2024 Dec;61(12):1981-1990. doi: 10.1177/10556656231190046. Epub 2023 Jul 24. PMID 37488938
- [Result] Behrens B, Swetlitz C, Pine DS, Pagliaccio D. The Screen for Child Anxiety Related Emotional Disorders (SCARED): Informant Discrepancy, Measurement Invariance, and Test-Retest Reliability. Child Psychiatry Hum Dev. 2019 Jun;50(3):473-482. doi: 10.1007/s10578-018-0854-0. PMID 30460424
- [Result] Peng, W., Yongjing, H., Likun, Z., Weiqi, Y., Xinrui, T., Fengyan, L., & Jihua, W. (2022). Evaluation of efficacy of expansion method for auricular reconstruction and quality of life in children with microtia. CHINESE JOURNAL OF AESTHETIC AND PLASTIC SURGERY, 33(4), 204-208. https://doi.org/https://doi.org/10.3969/j.issn.1673-7040.2022.04.004
- [Result] Ren YY, Zhao SQ. [Development and evaluation of a quality of life scale specific to patients with congenital external and middle ear malformation]. Zhonghua Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2010 Aug;45(8):623-7. Chinese. PMID 21055235
- [Result] Pickering PM, Osmotherly PG, Attia JR, McElduff P. An examination of outcome measures for pain and dysfunction in the cervical spine: a factor analysis. Spine (Phila Pa 1976). 2011 Apr 1;36(7):581-8. doi: 10.1097/BRS.0b013e3181d762da. PMID 21079542
- [Result] Dunstan DA, Scott N, Todd AK. Screening for anxiety and depression: reassessing the utility of the Zung scales. BMC Psychiatry. 2017 Sep 8;17(1):329. doi: 10.1186/s12888-017-1489-6. PMID 28886698